CLINICAL TRIAL: NCT05013073
Title: Adapting the ASTHMAxcel ED Application to Improve Asthma Related Patient-Centered Outcomes and Health Care Resource Utilization
Brief Title: ASTHMAXcel Emergency Department Study
Acronym: ASTHMAXcel
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB approval expired
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-12692
Record Dates: First submitted 2021-08-06; First posted 2021-08-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Asthma; Asthma Attack
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Single arm prospective open label study
Masking Description: Open Label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): All patients will be enrolled in a single arm and download the mobile application ASTHMAxcel ED to their smartphones.
  Interventions: Other: ASTHMAXcel ED Application

INTERVENTIONS:
Other: ASTHMAXcel ED Application — A mobile application designed to assist patients in asthma symptom recognition, treatment best practices, and trigger identification.

SUMMARY:
This protocol focuses on Phase 1 of a planned two-phase research project. Phase 1 aims to test and adapt a prototype ASTHMAXcelED application for the ED. Phase 2 will be an RCT to test the efficacy of a refined ASTHMAXcelED app after being modified based on the results of Phase 1.

DETAILED DESCRIPTION:
The original ASTHMAxcel app was developed by Dr. Jariwala, which delivers asthma education and promotes patients' adherence to the national asthma guidelines. The app was developed in accordance with Montefiore Medical Center's regulatory/compliance (determined by the Montefiore Legal department and Einstein-Montefiore Office of Biotechnology) and security (determined by Montefiore IT) policies. Over the last several years the app has been iteratively improved based on patient feedback and has been shown to improve asthma knowledge, asthma control, and asthma-related quality of life among asthma clinic patients. This version of the app has been tailored to the ED, requiring less physician directed education and focusing on common triggers and symptom management. Research associates will ask each patient to download the ASTHMAXcelED app and RA's instruct them on use of the application. RA's will also show every patient a video using the ASTHMAXcelED mobile application in which the investigators demonstrate correct use of an inhaler and discuss asthma triggers.

ELIGIBILITY:
Inclusion Criteria:

* English speakers
* at least 18+ years old with
* physician-diagnosed asthma.

Exclusion Criteria:

* severe cognitive or psychiatric conditions precluding capacity to provide informed consent,
* inability to speak English,
* lacking the technology to access the app.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test (ACT) | 4 Week Period
  A patient self-administered tool for identifying those with poorly controlled asthma.

SECONDARY OUTCOMES:
mini Asthma Quality of Life Questionnaire (mini AQLQ) | Recall over 2 week period
  Based on the 32 item AQLQ, the mini AQLQ is a 15-item self-administered tool constructed to meet the efficiency needs of large-scale clinical trials. The instrument was constructed for adults, and shown to have good reliability, responsiveness, construct and criterion validity. It captures functional impairments most relevant to adult asthma patients over a 2 week recall period. The tool is scored on a 7 point Likert scale, with increasing values corresponding with worsening quality of life.
Unified Theory of Acceptance and use of Technology | Measured at 4 weeks after intervention
  UTAUT explains user intention and behavior regarding the adoption of new technology. It explains user interaction using 4 domains: 1) performance expectancy, 2) effort expectancy, 3) social influence, and 4) facilitating conditions. The model explained 70% of the variance in Behavioral Intention to Use (BI) and about 50% in actual use, and has been validated against eight similar models and across nine culturally diverse nations.

OTHER OUTCOMES:
Open Ended Questions for ASTHMAXcelED Application Improvement | Measured at 4 weeks after intervention
  In order to iteratively improve the app and develop themes regarding user adoption, participants will be asked the following open ended questions and their answers transcribed in their entirety.
  How do you feel about using the app? Have you run into any issues using the app? Is it getting easier/harder to use the app over time? Which app features do you like? Which app features do you dislike? Which app features do you find difficult to use? How can the app be improved?

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Friedman, MD, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Montefiore Medical Center, Weiler Campus, The Bronx, New York
  - Montefiore Medical Center, Moses Campus, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rui, P., & Kang, K. (2014). National Hospital Ambulatory Medical Care Survey: 2014 Emergency Department Summary Tables. Retrieved from http://www.cdc.gov/nchs /data/ahcd/nhamcs_emergency/2014 _ed_web_tables.pdf
- [Background] Gerald JK, Denninghoff KR. Emergency Department Recidivism and Asthma: Revisiting an Old Problem. J Allergy Clin Immunol Pract. 2018 Nov-Dec;6(6):1914-1915. doi: 10.1016/j.jaip.2018.06.006. No abstract available. PMID 30390904
- [Background] Camargo CA Jr, Rachelefsky G, Schatz M. Managing asthma exacerbations in the emergency department: summary of the National Asthma Education And Prevention Program Expert Panel Report 3 guidelines for the management of asthma exacerbations. Proc Am Thorac Soc. 2009 Aug 1;6(4):357-66. doi: 10.1513/pats.P09ST2. No abstract available. PMID 19675345
- [Background] Hsia BC, Wu S, Mowrey WB, Jariwala SP. Evaluating the ASTHMAXcel Mobile Application Regarding Asthma Knowledge and Clinical Outcomes. Respir Care. 2020 Aug;65(8):1112-1119. doi: 10.4187/respcare.07550. Epub 2020 Jun 2. PMID 32487751
- [Background] "Asthma Control Test." Asthma Control Test (ACT), American Thoracic Society, www.thoracic.org/members/assemblies/assemblies/srn/questionaires/act.php
- [Background] Juniper EF, Guyatt GH, Cox FM, Ferrie PJ, King DR. Development and validation of the Mini Asthma Quality of Life Questionnaire. Eur Respir J. 1999 Jul;14(1):32-8. doi: 10.1034/j.1399-3003.1999.14a08.x. PMID 10489826
- [Background] Oshlyansky, Lidia, Paul Cairns, and Harold Thimbleby.